CLINICAL TRIAL: NCT07147647
Title: Efficacy of Direct Selective Laser Trabeculoplasty (DSLT) for Reducing Intraocular Pressure in Non-Caucasian Open Angle Glaucoma Patients
Brief Title: Direct Selective Laser Trabeculoplasty (DSLT) for Reducing Eye Pressure in Non-Caucasian Patients With Open Angle Glaucoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Select Eye Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-SG27
Record Dates: First submitted 2025-08-11; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Primary Open Angle Glaucoma (POAG)
Keywords: Direct Selective Laser Trabeculoplasty; DSLT; Primary Open Angle Glaucoma; POAG; Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Intervention Model Description: Prospective, Single-Arm, Open-Label Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Direct Selective Laser Trabeculoplasty (Experimental)
  Interventions: Device: Direct Selective Laser Trabeculoplasty

INTERVENTIONS:
Device: Direct Selective Laser Trabeculoplasty — DSLT using the Belkin Vision Eagle Device

SUMMARY:
The goal of this clinical trial is to to evaluate how well Direct Selective Laser Trabeculoplasty (DSLT) lowers eye pressure in eyes of adult, non-Caucasian participants with primary open angle glaucoma. The main question it aims to answer is:

What is the washed out eye pressure (eye pressure when not on any glaucoma medications) of participants 6 months after the Direct Selective Laser Trabeculoplasty (DSLT) procedure compared to the washed out eye pressure of participants prior to the DSLT procedure.

Participants will:

Undergo the DSLT procedure in one or both eyes and visit the clinic 1 month, 3 months, and 6 months after the procedure to have their vision and eye pressure measured.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate intraocular pressure (IOP) reduction of Direct Selective Laser Trabeculoplasty (DSLT) treatment in eyes of non-Caucasian patients with primary open angle glaucoma by assessing the washed out IOP reduction of DSLT at 6 months (compared to washed out baseline IOP), measuring the success rate of achieving ≥ to 20% IOP reduction from washed out baseline, assessing the proportion of medication-free eyes at 6 months post-DSLT, the need for secondary intervention (additional medications or procedures) at 6 months post-DSLT, and by comparing the washed out IOP reduction at 6 months post-DSLT compared to the washed out baseline IOP according to trabecular meshwork pigmentation grade.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of Black African descent scheduled to undergo DSLT treatment in one or both eyes.
* Diagnosis of mild to moderate primary open angle glaucoma (POAG).
* Mild to moderate POAG will be defined as Stage 2 or better of the Hodapp-Anderson-Parrish glaucoma staging system.
* Treatment naive or washed out IOP at time 0 ranging from ≥ 21 through 32 mm Hg.

Exclusion Criteria:

* Screened patients who were on IOP-lowering medications who did not successfully complete medication washout at the time of the procedure (time 0).
* Previous glaucoma surgeries/interventions:
* Patients who have undergone prior glaucoma-related procedures (e.g., trabeculectomy, laser trabeculoplasty, MIGS, or tube shunt).
* Secondary glaucoma:
* Patients with secondary forms of glaucoma, such as angle-closure glaucoma, neovascular glaucoma, or glaucoma resulting from trauma or other systemic diseases.
* Other significant ocular conditions including advanced cataracts, retinal diseases (e.g., age-related macular degeneration), or any condition that might complicate the assessment of intraocular pressure (IOP) or visual function as deemed by the investigator.
* Subjects who are pregnant, breast-feeding, or intend to become pregnant during the study period as determined by verbal inquiry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
IOP reduction at 6 months washed out post-DSLT compared with washed out baseline IOP. | 6 Months post-DSLT

SECONDARY OUTCOMES:
Proportion of eyes with ≥ 20% washed out IOP reduction at 6 months post-DSLT without secondary interventions (additional medications or procedures) compared with washed out baseline IOP. | 6 months post-DSLT
Proportion of medication free eyes at 6 months post-DSLT | 6 Months Post-DSLT
  Eyes not using any glaucoma medications
The number of participants who require secondary interventions (additional IOP-lowering procedures) prior to the completion of the 6 month post-DSLT visit. | 6 Months Post-DSLT
The number of participants who require secondary interventions (additional IOP-lowering medications) prior to the completion of the 6 month post-DSLT visit. | 6 Months Post-DSLT
Change in 1 month and 3 month non-washed out IOP vs washed out baseline IOP | 1 month and 3 months post-DSLT
  Measured in mmHg by Goldmann Applanation Tonometry
Mean 6 month washed out IOP reduction compared with washed out baseline IOP stratified by Trabecular Meshwork pigmentation grade. | 6 Month Post-DSLT
  Trabecular meshwork pigment will be graded on a scale of 0-4 where 0 is no pigment and 4 is heavy pigmentation

CONTACTS AND LOCATIONS:
Locations (1):
- Select Eye Care, Elkridge, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Not applicable; individual participant-level data will not be shared

REFERENCES:
- [Background] Gafvels M, Bengtsson-Olivecrona G, Olivecrona T. Correlation of plasma progesterone concentrations to ovarian H-type lipase activity during pseudopregnancy in the rat. J Reprod Fertil. 1989 Jul;86(2):589-98. doi: 10.1530/jrf.0.0860589. PMID 2760888
- [Background] Mills RP, Budenz DL, Lee PP, Noecker RJ, Walt JG, Siegartel LR, Evans SJ, Doyle JJ. Categorizing the stage of glaucoma from pre-diagnosis to end-stage disease. Am J Ophthalmol. 2006 Jan;141(1):24-30. doi: 10.1016/j.ajo.2005.07.044. PMID 16386972
- [Background] Hughes BA, Bacharach J, Craven ER, Kaback MB, Mallick S, Landry TA, Bergamini MV. A three-month, multicenter, double-masked study of the safety and efficacy of travoprost 0.004%/timolol 0.5% ophthalmic solution compared to travoprost 0.004% ophthalmic solution and timolol 0.5% dosed concomitantly in subjects with open angle glaucoma or ocular hypertension. J Glaucoma. 2005 Oct;14(5):392-9. doi: 10.1097/01.ijg.0000176935.08392.14. PMID 16148589
- [Background] Racette L, Wilson MR, Zangwill LM, Weinreb RN, Sample PA. Primary open-angle glaucoma in blacks: a review. Surv Ophthalmol. 2003 May-Jun;48(3):295-313. doi: 10.1016/s0039-6257(03)00028-6. PMID 12745004
- [Background] Kass MA, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Gordon MO. The Ocular Hypertension Treatment Study: a randomized trial determines that topical ocular hypotensive medication delays or prevents the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):701-13; discussion 829-30. doi: 10.1001/archopht.120.6.701. PMID 12049574
- [Background] Gazzard G, Konstantakopoulou E, Garway-Heath D, Adeleke M, Vickerstaff V, Ambler G, Hunter R, Bunce C, Nathwani N, Barton K; LiGHT Trial Study Group. Laser in Glaucoma and Ocular Hypertension (LiGHT) Trial: Six-Year Results of Primary Selective Laser Trabeculoplasty versus Eye Drops for the Treatment of Glaucoma and Ocular Hypertension. Ophthalmology. 2023 Feb;130(2):139-151. doi: 10.1016/j.ophtha.2022.09.009. Epub 2022 Sep 17. PMID 36122660
- [Background] Congdon N, Azuara-Blanco A, Solberg Y, Traverso CE, Iester M, Cutolo CA, Bagnis A, Aung T, Fudemberg SJ, Lindstrom R, Samuelson T, Singh K, Blumenthal EZ, Gazzard G; GLAUrious study group. Direct selective laser trabeculoplasty in open angle glaucoma study design: a multicentre, randomised, controlled, investigator-masked trial (GLAUrious). Br J Ophthalmol. 2023 Jan;107(1):62-65. doi: 10.1136/bjophthalmol-2021-319379. Epub 2021 Aug 25. PMID 34433548
- [Background] Goldenfeld M, Belkin M, Dobkin-Bekman M, Sacks Z, Blum Meirovitch S, Geffen N, Leshno A, Skaat A. Automated Direct Selective Laser Trabeculoplasty: First Prospective Clinical Trial. Transl Vis Sci Technol. 2021 Mar 1;10(3):5. doi: 10.1167/tvst.10.3.5. PMID 34003939
- See also: Change in Intraocular Pressure after Selective Laser Trabeculoplasty in North Indian Primary Open Angle Glaucoma Patients: A Prospective Analytical Study — https://doi.org/10.7860/JCDR/2024/74217.20250